CLINICAL TRIAL: NCT01129765
Title: Home Usability of a Nasal Lavage System in Children
Status: Completed | Type: Observational
Sponsor: Aardvark Medical Company (Industry)
Responsible Party: Richard Schwartz, MD, Advanced Pediatrics
Other Study IDs: AM-002
Record Dates: First submitted 2010-05-21; First posted 2010-05-25 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Nasal Congestion; Respiratory Tract Infection; Sinusitis; Allergic Rhinitis
Keywords: Nasal suction; Nasal aspiration; Nasal saline irrigation; Nasal lavage
MeSH Terms: conditions — Nasal Obstruction; Respiratory Tract Infections; Sinusitis; Rhinitis, Allergic | interventions — Nasal Lavage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parents of congested children: Parents of children less than six years of age with nasal congestion for which nasal suctioning and salt water irrigation is traditionally recommended.
  Interventions: Device: Use of an automatic nasal irrigator/aspirator

INTERVENTIONS:
Device: Use of an automatic nasal irrigator/aspirator — After reading the device's user manual, parents were asked to use it on their congested children to their satisfaction. During this time, a clinical observer recorded predetermined steps that needed to be performed for success as well as presence of any adverse events.
  Other Names: Nasal aspiration; Nasal irrigation; Nasal lavage

SUMMARY:
This study evaluates labeling comprehension, ease of use and effectiveness of a new device for nasal and sinus irrigation and/or aspiration. The device is currently cleared for professional use and home use with a prescription. This is a usability study to demonstrate that this device is appropriate for home use.

DETAILED DESCRIPTION:
Nasal congestion is an important complication of viral upper respiratory infections in young children. It can lead to poor eating, sleeping and breathing. Recently, the FDA recommended against using over-the-counter cold remedies in young children because of inefficacy and occasional dangerous side effects. A commonly recommended non-drug solution for nasal congestion is nasal suctioning. This can be effective but currently available methods have been found to be awkward, uncomfortable and ineffective.

The studied device has potential for making nasal suctioning easy to perform in the home setting, especially in young children. It is already FDA cleared for professional use and this study was developed to demonstrate that it is appropriate for the home as well. This would be significant as it would allow parents a strategy of clearing their child's nose without drugs.

The device is automatic and handheld that can irrigate and/or aspirate the nasal cavity with hospital-grade suction. The handle houses a pump that can achieve air flows known to be effective for infant nasal suctioning in the hospital. A disposable wash-head is placed on top. It has an irrigation chamber with 0.9% saline and another chamber for collecting the aspirated nasal contents. The unit operates from a single bi-functional button.

Several key safety features have been built in such as: a tip that is shaped to maximize the seal but prevent intrusion into the nose; an irrigation function that delivers an optimal volume but prevents flooding the nasal cavity; and a pump that can deliver suction known to be effective in the hospital but whose safety valve does not allow it to rise above dangerous levels.

Participants were parents of children who have nasal congestion for whom nasal suctioning is traditionally recommended. They were asked to review the instruction manual of the device, and then use it on their children.

The primary outcome was proper use of device that was precisely defined. Additionally, subjective efficacy of mucus removal, evidence of adverse events and understanding of the device's user manual were also measured.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children less than 6 years of age who were suffering from nasal congestion for which nasal suctioning and salt water irrigation/drops are prescribed.

Exclusion Criteria:

* Parents of children in marked respiratory distress or who maxillofacial malformations not conducive to nasal suctioning.
* Additionally, parents of children with recurrent nose bleeds, bleeding disorders or irritated peri-nasal skin were excluded.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The participants were selected from a primary care pediatric clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schwartz, MD, Principal Investigator — Advanced Pediatrics
Locations (1):
- Advanced Pediatrics, Vienna, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in a pediatric ambulatory clinic in July and August of 2009. The clinical coordinator identified patients as they presented to the clinic if they met inclusion criteria and informed consent was obtained before patient entry.
Period: Overall Study
Arm/Group | Parents of Congested Children
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Parents of Congested Children
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.75 (0.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Experienced Ease of Use With the Device
Description: After using the device, the caregiver answered this question on a five point Likert-like scale with increasing favorability with increasing number. An answer of 3 or greater is considered an affirmative answer. Such responses reported along with the exact 95% confidence intervals.
  The question and scale are as follows: How easy was the device to use?
  1 difficult, 2 somewhat hard, 3 fairly easy, 4 easy, 5 very easy
Time Frame: Day one, immediately
Population: This was the total number of participants who answered this question.
Measure: Number; unit: participants
Arm/Group | Parents of Congested Children
Number analyzed (Participants) | 30
participants | 29
Statistical Analysis 1: Comparison: Parents of Congested Children; Proportion responding >=3 on a 5-point likert scale, with exact 95% confidence interval from the binomial distribution; Test type: Superiority or Other; Descriptive; Proportion = 0.97, 95% CI 2-sided [0.83 to 1.0]

2. Secondary Outcome: Number of Participants Who Found the Device to be Effective
Description: After using the device, the caregiver answered this question on a five point Likert-like scale with increasing favorability with increasing number. The proportion answering 3 or greater is reported along with the exact 95% confidence intervals.
  The question and scale are as follows: How well did the device remove nasal secretions?
  1 difficult, 2 somewhat hard, 3 fairly easy, 4 easy, 5 very easy
Time Frame: Day one, immediately
Measure: Number; unit: participants
Arm/Group | Parents of Congested Children
Number analyzed (Participants) | 30
participants | 29
Statistical Analysis 1: Comparison: Parents of Congested Children; Descriptive summary of proportion responding >=3 on 5-point Likert scale, with exact 95% confidnce interval from the binomial distribution; Test type: Superiority or Other; Descriptive; Proportion = 0.97, 95% CI 2-sided [0.83 to 1.0]

3. Primary Outcome: Number of Participants Who Properly Used the Nasal Irrigator/Aspirator Device
Description: 'Proper use' is defined as successfully completing all of the following five steps:
  1. Attaching wash-head to handle properly
  2. Positioning child correctly for procedure as per the user manual's instructions
  3. Using the device's control button correctly for both irrigation and aspiration
  4. Placing the wash-head tip correctly at the nasal opening
  5. Using the device for up to but not exceeding five seconds
Time Frame: Day one, immediately
Measure: Number; unit: participants
Arm/Group | Parents of Congested Children
Number analyzed (Participants) | 30
participants | 29 [83% to 100%]
Statistical Analysis 1: Comparison: Parents of Congested Children; Null hypothesis: Pr ≤ 0.7 versus HA: Pr > 0.7; Pr is proportion using device appropriately. Observed rate calculated with exact 95% confidence interval from the binomial distribution. 2-sided p-value from binomial distribution. With the proposed sample size of 30 subjects, we will reject the primary null hypothesis if at least 27 are observed to use the device properly. We will have 80% power for this to occur provided that the true rate in the population is at least 92%; Test type: Superiority or Other; p = 0.0005, One-sample proportion; Proportion = 0.97, 95% CI 2-sided [0.83 to 1.0]

4. Secondary Outcome: Number of Participants Who Identified the Device's User Manual as Easy to Understand
Description: After using the device, the caregiver answered this question on a five point Likert-like scale with increasing favorability with increasing number. The proportion answering 3 or greater is reported along with the exact 95% confidence intervals.
  The question and scale are as follows: How easy was the manual to understand?
  1 difficult, 2 somewhat hard, 3 fairly easy, 4 easy, 5 very easy
Time Frame: Day one, immediately
Measure: Number; unit: participants
Arm/Group | Parents of Congested Children
Number analyzed (Participants) | 30
participants | 30
Statistical Analysis 1: Comparison: Parents of Congested Children; Descriptive summary of proportion responding >=3 on a 5-point Likert scale, with exact 95% confidnce interval from the binomial distribution; Test type: Superiority or Other; Descriptive; Proportion = 1.0, 95% CI 2-sided [0.88 to 1.0]

5. Secondary Outcome: Number of Patients Who Were Observed to Have an Adverse Event
Description: While using the device, the patients were observed by the research coordinator for any of the following adverse events to occur:
  1. bloody nose
  2. being sprayed in the eye with the saline
  3. vomiting after the procedure
  4. choking during or after the procedure
  5. other
Time Frame: Day one, immediately
Measure: Number; unit: patients with an adverse event
Arm/Group | Parents of Congested Children
Number analyzed (Participants) | 30
patients with an adverse event | 0
Statistical Analysis 1: Comparison: Parents of Congested Children; Descriptive summary of proportion observed to have a safety issue, with exact 95% confidnce interval from the binomial distribution; Test type: Superiority or Other; Descriptive; Proportion = 0, 95% CI 2-sided [0 to 0.12]

6. Secondary Outcome: Number of Patients Experiencing a Physical Injury During Use
Description: After the procedure, the patient was directly examined for any of the following:
  1. bleeding from the nostrils
  2. disruption of the skin around the nose
  3. increased work of breathing/respiratory distress (increased respiratory rate, increased respiratory accessory muscle use)
Time Frame: Day one, immediately
Population: This is the total number of participants, all of whose children were examined after the procedure.
Measure: Number; unit: paricipants
Arm/Group | Parents of Congested Children
Number analyzed (Participants) | 30
paricipants | 0
Statistical Analysis 1: Comparison: Parents of Congested Children; Descriptive summary of proportion found to have injury, with exact 95% confidnce interval from the binomial distribution; Test type: Superiority or Other; Descriptive; Proportion = 0, 95% CI 2-sided [0 to 0.12]

ADVERSE EVENTS:
Arm/Group | Parents of Congested Children
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No